CLINICAL TRIAL: NCT01965977
Title: Open-label, Multicenter Phase II Study of Bortezomib for Maintenance Therapy in Patients With High Risk Diffuse Large B Cell Lymphoma
Brief Title: Bortezomib Maintenance in High Risk DLBCL
Acronym: Borma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Won Seog Kim, MD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SMC2013-04-124
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): bortezomib 1.3mg/m2 subcutaneous on day 1 and15
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3mg/m2, on day 1 and 15 SC Repeat every month for 12months
  Other Names: velcade

SUMMARY:
This study is an Open-labeled, multicenter Phase II study of Bortezomib for maintenance therapy in patients with high risk diffuse large B cell lymphoma (DLBCL). Primary objective is 3 years relapse free survival (RFS) and Secondary objectives are 3 years overall survival (OS), 3 years event free survival (EFS),Toxicities profiles, Quality of Life (FACT&GOG-Ntx)

DETAILED DESCRIPTION:
High-intermediate or high risk in IPI has a long-term chance of cure in the range about 50% in patients with DLBCL treated by R-CHOP. These high risk patients should be considered for additional new treatment to standard R-CHOP or investigational approaches in the context of clinical trials that are designed to ensure that potentially curative therapy.

Bortezomib has shown activity in vitro against DLBCL-derived cell lines. Single-agent bortezomib or chemotherapy combined bortezomib are feasible in follicular, mantle cell, marginal zone lymphoma and DLBCL with manageable toxicities. Bortezomib enhances the activity of chemotherapy in non-GCB but not GCB DLBCL, and provide a rational therapeutic approach based on genetically distinct DLBCL subtypes.

High CR/CRu rate with bortezomib with standard R-CHOP suggests it may be a good backbone for additional maintenance leading to durable response. However, there is no study of bortezomib as maintenance therapy after treated with R-CHOP in high risk patients with DLBCL. So we applied additional bortezomib as maintenance therapy in order to assess improving efficacy and survival rates in high risk patients with non-GCB DLBCL who had been confirmed CR after treated with R-CHOP.

ELIGIBILITY:
Inclusion Criteria:

1. Newly histologically confirmed CD20 positive diffuse large B-cell lymphomas and only Non-GCB type will be included
2. High intermediate or high risk by IPI risk, or Bulky mass ≥ 10cm at diagnosis
3. Complete response is confirmed after six or eight cycles R-CHOP chemotherapy by CT scan with confirmed negative PET-CT based on the Revised International Workshop Criteria.
4. Additional surgery or radiotherapy are accepted
5. Age ≥ 20
6. Performance status (ECOG) ≤ 2
7. Adeqaute renal function: Cr < 2.5 mg/dL
8. Adeqaute liver functions: Transaminase (AST/ALT) < 3 x upper normal value UNV)Bilirubin < 1.5 x UNV Alkaline phosphatase < 5 xUNV
9. Adeqaute BM functions: ANC > 1,000/uL and platelet > 75,000/uL and hemoglobin > 9.0 g/dL
10. Written Informed consent

Exclusion Criteria:

1. Tumor response after 6-8 cycles CTx< CR
2. Consider stem cell transplantation
3. Central nervous system (CNS) metastases
4. Pregnant or lactating women, patients of childbearing potential not employing adequate contraception
5. Other serious illness or medical conditions A. Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry B. History of significant neurologic or psychiatric disorders including dementia or seizures C. Active uncontrolled infection
6. Any other malignancies within the past 5 years except curatively treated non- melanoma skin cancer or in situ carcinoma of cervix uteri.
7. Prior history of allegic reaction to study treatment drugs
8. Peripheral neuropathy grade 2 or worse
9. DLBCL of the testis and primary mediastinal DLBCL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
3years relapse free survival | from the date of first drug administration until the date of last follow up, assessed up to 4years
  3years relapse free survival will be assessed after starting maintenance therapy for 1year and then following up for 3years.

SECONDARY OUTCOMES:
3years overall survival | from the date of first drug administration until the date of last follow up, assessed up to 4years
  3years overall survival will be assessed after starting maintenance therapy for 1year and then following up for 3years.
3years event free survival | from the date of first drug administration until the date of last follow up, assessed up to 4years
  3years event free survival will be assessed after starting maintenance therapy for 1year and then following up for 3years.
Toxicity profiles | from the date of first drug administration until the date of the 30th day after last cycle of chemotherapy
  Safety profiles will be evaluated using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Quality of life scale | from the date of first drug administration until the date of last follow up, assessed up to 4years
  Quality of life will be assessed after starting maintenance therapy for 1year and then following up for 3years by using FACT&GOG-Ntx.

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea